CLINICAL TRIAL: NCT05201950
Title: Pilot Randomised Controlled Trial of Virtual Patient Simulation Versus In-situ Simulation for Improving Performance in Trauma and Sepsis Resuscitation in Junior Clinicians in the Emergency Department
Brief Title: Study of Virtual Simulated Resuscitation in Junior Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DSRB 2021/00542
Record Dates: First submitted 2021-12-16; First posted 2022-01-21 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-01

CONDITIONS: Education, Medical

STUDY DESIGN:
Intervention Model Description: Participants are assigned to learning through either virtual simulation, or team based in situ simulation, and are not planned to cross over during the study period.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants: it is not feasible to mask participants from their educational intervention Investigator: Two investigators (JCL and LZY) will not be masked as they will be scheduling and delivering interventions. The remaining investigators will be masked, including those assisting participants as standardised assistants during outcome assessment simulation.
  Outcome assessors: They will be masked from participants' group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual simulation (Experimental): - Virtual simulation group: Participants will log in to the virtual simulation software from home and play 2 cases (1 case of sepsis, 1 case of trauma). Learners are instructed to play each case as many times as they like within 70 minutes, to reach the highest score possible in that time. This process is proctored, with participants sharing their screen over video conferencing with study team members (JCL or LZY) to ensure adherence to time limit and cases played.
  Interventions: Other: Virtual simulation
- Team based in situ simulation (Active Comparator): - Team based in situ simulation group: Faculty observing and debriefing learners at the mock code will be variable and consist of a wide range of NUH emergency department faculty outside of this study, due to logistical constraints in having the same faculty being present consistently in the entire year. The in situ simulation will cover 1 case of sepsis, and 1 case of trauma, with case content matched to the cases in the virtual simulation group, and time matched at 70 minutes.
  Interventions: Other: Team based in situ simulation

INTERVENTIONS:
Other: Virtual simulation — Virtual simulation using Full-Code, a virtual simulation software with a bank of emergency medicine cases
  Arms: Virtual simulation
Other: Team based in situ simulation — In situ simulation, using a high fidelity manikin in the critical care area of the emergency department, with team members consisting of multiple junior doctors and nurses, facilitated by senior emergency medicine doctors and nurses.
  Arms: Team based in situ simulation

SUMMARY:
The investigators seek to examine the impact of virtual patient simulation on junior clinicians' resuscitation skills in an academic emergency department.

Exposure to real life resuscitation cases is opportunistic, with variation in case mix across different junior clinicians. Junior clinicians are closely supervised during resuscitations, with limited independence to make decisions, for patient safety.

High fidelity simulation, such as in-situ mock codes with a high fidelity manikin, is resource intensive. Constraints in facilitator and learner time and manpower reduce the feasibility of holding large numbers of simulations for large numbers of learners, leading to limited breadth of case mix exposure in simulation cases.

Virtual patient simulation may allow greater and more uniform breadth of exposure and allow automated feedback and rapid cycle deliberate practiceacross a wide range of cases, with reduced resource intensiveness, and prepare them to better utilise limited opportunities for resuscitation during real life or high fidelity simulation.

Virtual simulators have been found to be useful for improving skills rather than knowledge or attitudes in health professions education. Such skills include communication, radiograph interpretation, dermatological diagnosis, and cardiac arrest procedures.

What is not known is:

1. Whether going directly to in-situ simulation with a high fidelity manikin is the best learning approach for resuscitation, given its potentially detrimental high cognitive load, compared to going first to virtual patient simulation.
2. Whether the benefits of virtual simulation extend beyond cardiac arrest and to other resuscitation scenarios, such as trauma, sepsis, and others.

The investigators' hypothesis is that in junior clinicians in the emergency department who have received didactic materials in trauma and sepsis resuscitation, proceeding next to learning by virtual patient resuscitation simulation is associated with improved scores in resuscitation performance for trauma and sepsis, as measured by checklists of required actions during observed in-situ simulation with a high-fidelity manikin, compared to proceeding next to learning by team-based in-situ simulation with a high fidelity manikin. This pilot study aims to determine the feasibility of a randomised controlled trial to test the above hypothesis.

DETAILED DESCRIPTION:
Sample size: For a pilot study, a sample size of at 24-50 participants is advisable to be informative regarding population characteristics such as expected means and standard deviation, to facilitate future study, where sample size calculation will target a small standardised effect size of 0.2, where standardised effect size would be the difference in means divided by standard deviation. About 50 junior clinicians are anticipated to rotate through NUH emergency department for at least 3 months in 2022.

Randomisation:

- After informed consent and recruitment, participants will be randomised to virtual simulation versus in-situ simulation groups, through the use of opaque sealed envelopes. The randomisation sequence will be generated by one investigator (A), with block randomisation in varying block sizes, while another investigator (B) will open envelopes to allocate learners to their groups, to maintain allocation concealment.

Interventions:

* Two investigators (C and D) will schedule participants for assigned interventions, namely virtual simulation or team-based in-situ simulation. As team-based in-situ simulation sessions are dispersed across each month, virtual simulation sessions will be matched to in-situ simulation days, to prevent confounding by time from outcome assessment. All interventions will be scheduled after didactic materials for resuscitation have been delivered to learners as part of standard departmental curriculum.
* Virtual simulation group: Participants will log in to the virtual simulation software from home and play 2 cases (1 case of sepsis, 1 case of trauma). Participants are instructed to play each case as many times as personally desired within 70 minutes, to reach the highest score possible in that time. This process is proctored, with participants sharing their screen over video conferencing with two investigators (C and D) to ensure adherence to time limit and cases played.
* Team based in situ simulation group: Faculty observing and debriefing learners at the mock code will be variable and consist of a wide range of NUH emergency department faculty outside of this study, due to logistical constraints in having the same faculty being present consistently in the entire year. The in situ simulation will cover 1 case of sepsis, and 1 case of trauma, with case content matched to the cases in the virtual simulation group, and time matched at 70 minutes.

Outcome assessment:

* Scores obtained based on number of correct actions completed in a timely manner, during simulated resuscitation with a high fidelity manikin around the end of the 3rd month of their posting, as compared to a checklist of required actions derived from expert consensus among NUH emergency department clinicians, and aligned to established international guidelines for resuscitation in sepsis or trauma (e.g. Advanced Trauma Life Support 10th edition).
* Two trained and standardised assistants, playing the roles of one nurse and one doctor, will be present to assist the medical officer, who will take the role of resuscitation team leader.
* Each study participant will be observed and marked on two scenarios: one scenario on major trauma resuscitation, and one scenario on resuscitation of a patient with sepsis. Marking will be performed independently by two investigators (E and F) who will calibrate and standardise their ratings by watching one investigator (A) perform simulated resuscitation at different levels of competence, and using that as a stimulus to calibrate their ratings.
* All assistants and assessors doing marking will be blinded to participant allocation, and will not be involved in team based in situ simulated resuscitation during the study period.

Other data collection:

* Learner demographic data, level of post graduate experience generally and in emergency medicine, and views regarding assigned intervention (i.e. Kirkpatrick level of reaction), will be collected via an online questionnaire.
* The following virtual simulation metrics will be automatically captured: Number of attempts for each unique case, time spent on each attempt, scores obtained during each attempt as marked by a virtual patient simulator

Data analysis:

- Descriptive statistics of the following will be tabulated:

* Baseline characteristics of learners in each group, to determine effectiveness of randomisation
* Learner reaction data, to determine extent of acceptability of virtual patient simulation based on learner perception
* Mean, median, and measures of spread (either standard deviationor interquartile range, depending on whether data is normally distributed) of scores obtained

Analysis for associations:

* Primary outcome: Association between exposure to virtual patient simulation (categorical variable) and marks obtained during observed in-situ resuscitation using a high fidelity manikin (likely to be a continuous variable with normal distribution, and this pilot study would help to determine if that is true), as measured by number of correct actions completed on a checklist derived from local expert consensus, rated by two independent observers (Investigators E and F) with statistical testing using a 2-tailed student t-test.

  --> Interobserver agreement will be measured using intra class correlation
* The investigators acknowledge that as a pilot, the analyses are unlikely to be adequately powered. Nonetheless, understanding the distribution of marks in each group, including mean/median/measures of variance, would be useful for planning further study.

ELIGIBILITY:
Inclusion Criteria:

* Junior doctors scheduled to rotate through NUH emergency department for at least 3 months

Exclusion Criteria:

* Pregnant women will be excluded from the study as the study procedures do involve additional exposure to fellow healthcare workers, with the associated risk of COVID transmission, while there is no direct benefit in terms of generalisable knowledge about pregnancy or the fetus.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Score obtained in outcome assessment simulation | At end of 3rd month of junior clinicians' emergency medicine rotation
  Participants will be assessed by 2 independent assessors using a standardised checklist during simulation with a high fidelity manikin and standardised assistants in two scenarios: trauma, and sepsis

SECONDARY OUTCOMES:
Learner satisfaction | Within one week after completion of assigned intervention
  Participants report their level of satisfaction with the intervention through an online questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew JW Low, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Low MJW, Chan GWH, Li Z, Koh Y, Jen CL, Lee ZY, Cheng LTW. Comparison of virtual and in-person simulations for sepsis and trauma resuscitation training in Singapore: a randomized controlled trial. J Educ Eval Health Prof. 2024;21:33. doi: 10.3352/jeehp.2024.21.33. Epub 2024 Nov 18. PMID 39552082